CLINICAL TRIAL: NCT06212414
Title: Mind Programme for Women With Breast Cancer: A Randomized Controlled Trial Testing the Programme´s Cost-effectiveness and Efficacy in Changing Psychological and Biological Outcomes (Nationwide Coverage)
Brief Title: Mind Programme for Women With Breast Cancer (Nationwide Coverage)
Acronym: MIND(n)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Coimbra (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Inês A Trindade, Principal investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CINEICC-3-IAT(n)
Record Dates: First submitted 2024-01-03; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer Female
Keywords: Mental health; Quality of life; Cost-effectiveness; Mindfulness; Compassion Focused Therapy; Acceptance and Commitment Therapy
MeSH Terms: conditions — Psychological Well-Being | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mind programme (Experimental): This group will receive the Mind programme. This intervention comprises 8 weekly group sessions, with the duration of 120 minutes each, to be delivered via Zoom. Integration of Acceptance and Commitment Therapy, mindfulness and Compassion Focused Therapy components, adapted to women with breast cancer.
  All participants will continue on receiving the recommended medical treatment for their clinical diagnosis.
  Interventions: Behavioral: Mind Programme
- Support group (Active Comparator): This group will receive a 8-week support group intervention (weekly sessions, with the duration of 120 minutes each), via Zoom.
  All participants will continue on receiving the recommended medical treatment for their clinical diagnosis.
  Interventions: Behavioral: Support Group
- Waiting list (Treatment As Usual / No psychological intervention) (No Intervention): This group will receive the (psychological) treatment as usual in Portugal (no treatment), besides the recommended medical treatment for their clinical diagnosis. At the end of this research project, the intervention that proves to be most efficacious will be offered to participants from the waiting list condition.

INTERVENTIONS:
Behavioral: Mind Programme — Intervention based on Acceptance and Commitment Therapy, mindfulness, and compassion approaches
  Arms: Mind programme
Behavioral: Support Group — This intervention promotes the sharing of cancer-related experiences, active listening, and a sense of community between participants
  Arms: Support group

SUMMARY:
The purpose of this research project is to optimize the Mind programme for women with breast cancer, taking into consideration the results from its pilot study, and to testits efficacy and cost-effectiveness through a 3-arm randomized controlled trial

ELIGIBILITY:
Inclusion criteria:

1. age between 18-70;
2. primary diagnosis of BC (stages between I and III);
3. having a scheduled radiotherapy treatment starting within 2 months, currently undergoing radiotherapy treatment, or having finished radiotherapy treatment no more than 6 months prior, at any hospital in Portugal;
4. able to understand and answer to self-report questionnaires in Portuguese;
5. having access to a computer or tablet with internet.

Exclusion criteria:

1. currently undergoing any form of psychological intervention;
2. current diagnosis of severe psychiatric illness (psychotic disorder, bipolar disorder, substance abuse, and personality disorder) or suicidal ideation;
3. diagnosis of neurological disease.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline cancer-specific quality of life at post-treatment and 6-month follow-up | Baseline, post-treatment (2 months after baseline) and 6-month follow-up
  EORTC QLQ-C30

SECONDARY OUTCOMES:
Change from baseline depressive symptoms and anxiety severity at post-treatment and 6-month follow-up | Baseline, post-treatment (2 months after baseline) and 6-month follow-up
  Hospital Anxiety and Depression Scale
Change from baseline psychological flexibility at post-treatment and 6-month follow-up | Baseline, post-treatment (2 months after baseline) and 6-month follow-up
  Comprehensive Assessment of Acceptance and Commitment Therapy Processes
Change from baseline self-compassion and mindfulness at post-treatment and 6-month follow-up | Baseline, post-treatment (2 months after baseline) and 6-month follow-up
  Self-Compassion Scale
Change from baseline health-related quality of life at post-treatment and 6-month follow-up | Baseline, post-treatment (2 months after baseline) and 6-month follow-up
  EQ-5D-5L
Change from baseline consumption of resources and costs in breast cancer at post-treatment and 6-month follow-up | Baseline, post-treatment (2 months after baseline) and 6-month follow-up
  This questionnaire was developed by the research team and adapted from the UK Cancer Costs Questionnaire (UKCC) Version 2.0 to assess the consumption of resources and economic costs associated with breast cancer.
Major life events - controlling variable | 6-month follow-up
  Major Life Events Questionnaire
Sociodemographic and clinical variables - controlling variables | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Research in Neuropsychology and Cognitive and Behavioral Intervention, University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trindade IA, Soares A, Skvarc D, Carreiras D, Pereira J, Lourenco O, Sampaio F, de Sousa B, Martins TC, Boaventura P, Marta-Simoes J; Mind Project Team; Moreira H. Efficacy and cost-effectiveness of an ACT and compassion-based intervention for women with breast cancer: study protocol of two randomised controlled trials 1. Trials. 2025 Jan 3;26(1):5. doi: 10.1186/s13063-024-08626-4. PMID 39754194